CLINICAL TRIAL: NCT01628783
Title: Sequence Towards Remission in Depression
Acronym: STRIDE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jesper Ekelund (Other)
Collaborators: Academy of Finland (Other)
Responsible Party: Sponsor-Investigator, Jesper Ekelund, Professor of Psychiatry, University of Helsinki
Organization: University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-002476-14
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Depression
Keywords: Depression; emotional processing; fMRI; autobiographic memory; moderator of treatment response; mediator of treatment response
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Microgranular cellulose in gelatine capsules.
  Interventions: Drug: Placebo
- Escitalopram 10 mg (Experimental): Escitalopram in gelatine capsule
  Interventions: Drug: escitalopram 10 mg

INTERVENTIONS:
Drug: escitalopram 10 mg — orally once daily
  Arms: Escitalopram 10 mg
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
In this study the investigators use clinical, biological and imaging markers to develop predictive markers for remission from depression. The investigators compare individuals who have received placebo to individuals who have received 10 mg of escitalopram for one week. In this double-blind, randomized study the investigators a) compare the groups to observe the short-term effects of escitalopram and b) study the predictive value of these observations with respect to remission. Measures include, but are not restricted to, limbic emotional reactivity as assessed by fMRI, emotional processing, emotional memory, autobiographical memory.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder with current major depressive episode according to a SCID-I/P interview
* Montgomery-Åsberg depression rating score 15-30
* Age 18-60

Exclusion Criteria:

* Borderline, schizoid or schizotypal personality, bipolar or any psychotic disorder
* Primary diagnosis is anxiety disorder: 300.00, .01, .02, .21, .22, .29, .23, .3, 309.81, 308.3, 293.89
* Significant current suicidal ideation, or history of a suicide attempt
* Lifetime substance dependence; Last-year substance abuse; Last month over 24/16 standard doses of alcohol/week; Lifetime use of illicit substances > x5; Any illicit substance use in last month
* Depressive disorder due to medical condition or chemical substance
* Antidepressant medication use in last 4 months
* Severe, unstable somatic illness
* Use of antipsychotics, mood stabilizers, systemic corticosteroids, β-blockers or daytime benzodiazepines (a small dose of ≤10mg zolpidem once daily is permissible)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg rating scale | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erkki Isometsä, MD-PhD, Principal Investigator — University of Helsinki; Jesper Ekelund, MD-PhD, Principal Investigator — University of Helsinki
Locations (1):
- Helsinki University Central Hospital, Psychiatry Centre, Helsinki, Finland